CLINICAL TRIAL: NCT00225966
Title: Patient Registry to Study the Tined Lead Used With the InterStim System For Urinary Control
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study design was changed and is now InSite trial #1634 - See NCT00547378
Sponsor: MedtronicNeuro (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MGU-003
Record Dates: First submitted 2005-09-12; First posted 2005-09-26 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Urge Incontinence; Urinary Retention
Keywords: Urinary urgency-frequency
MeSH Terms: conditions — Urinary Incontinence, Urge; Urinary Retention

INTERVENTIONS:
Device: Device Medtronic InterStim Tined Leads Models 3889 and 3093

SUMMARY:
The purpose of this study is assess the long-term safety and effectiveness of the InterStim tined lead using a minimally invasive approach.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent
* 16 years of age or greater
* Willing and able to complete voiding diaries and questionnaires at various time points during the study
* Located geographically near the physician, or willing and able to travel to the physician's site as necessary for all required visits
* Failed or is not a candidate for more conservative treatment

Exclusion Criteria:

* Severe or uncontrolled diabetes; or diabetes with peripheral nerve involvement
* Pregnancy or planned pregnancy
* Concomitant medical conditions which would limit the success of the procedure such as: pelvic pain with uncertain etiology, active degenerative disc disease, spinal cord injury less than six months old, bleeding complications, or a cerebrovascular accident (CVA) less than six months old.
* Anatomical limitations that would prevent successful placement of an electrode
* Neurological diseases such as multiple sclerosis, clinically significant peripheral neuropathy or complete spinal cord injury (e.g., paraplegia)
* Subject characteristics indicating a poor understanding of the study or poor compliance with the study protocol (e.g. subjects with psychological and/or emotional problems, subjects unable to adequately operate equipment)
* Subjects with knowledge of planned magnetic resonance imaging (MRI), diathermy, microwave, high output ultrasonics, ultrasound scanning, or radiofrequency (RF) energy
* Mechanical obstruction such as benign prostatic hypertrophy, cancer, or urethral stricture
* Symptomatic urinary tract infection (UTI). Upon completion of therapy for UTI, or if the subject is receiving prophylaxis for UTI, subjects can be considered for test stimulation or the full system implant (whichever is applicable) if symptom free for one month prior to the procedure.
* Subjects with other implantable neurostimulators, pacemakers, or defibrillators
* Primary stress incontinence or mixed incontinence where the stress component overrides the urge component
* Active participation in another clinical study

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 153
Dates: Start 2004-08; Study Completion 2007-10

PRIMARY OUTCOMES:
Incidence of adverse events requiring surgical intervention
Incidence of lead migration

SECONDARY OUTCOMES:
Incidence of infection

CONTACTS AND LOCATIONS:
Overall Officials: Medtronic Investigator, Principal Investigator — Medtronic
Locations (2):
- United States (2):
  - Contact Medtronic for specific site information, Los Angeles, California
  - Contact Medtronic for site information, Minneapolis, Minnesota